CLINICAL TRIAL: NCT01351194
Title: Radiofrequency Ablation vs. Hepatic Resection for the Treatment of Hepatocellular Carcinomas Smaller Than 2 cm.A Prospective and Randomized Clinical Trial
Brief Title: Radiofrequency Ablation Versus Hepatic Resection for the Treatment of Hepatocellular Carcinomas Smaller Than 2 cm
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Cancer Center, Sun Yat-sen University, Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HCC0012
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2010-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; RFA; HR
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA group (Experimental): For PRFA, we used a commercially available system with a 375-KHz computer-assisted radiofrequency generator (Elektrotom HiTT 106, Berchtold, Medizinelektronik, Germany) and an open-perfused electrode (Berchtold, Tuttlingen, Germany) of 15 cm (or 20 cm), 14 Ga, and a 15 mm (or 20 mm) active electrode tip with microbores.
  Interventions: Procedure: RFA
- HR group (Experimental): SR was carried out under general anesthesia using a right subcostal incision with a midline extension. Intra-operative ultrasonography was performed routinely to evaluate the tumor burden, liver remnant, and the possibility of a negative resection margin. Anatomic resection, in the form of segmentectomy and/or subsegmentectomy as described by Makuuchi et al. (16) was the preferred surgical method of liver resection. Pringle's maneuver was routinely used with a clamp and unclamp time of 10 min and 5 min, respectively; this technique was used repeatedly throughout the entire procedure.
  Interventions: Procedure: hepatic resection

INTERVENTIONS:
Procedure: RFA — For PRFA, we used a commercially available system with a 375-KHz computer-assisted radiofrequency generator (Elektrotom HiTT 106, Berchtold, Medizinelektronik, Germany) and an open-perfused electrode (Berchtold, Tuttlingen, Germany) of 15 cm (or 20 cm), 14 Ga, and a 15 mm (or 20 mm) active electrode tip with microbores. The 14 Ga needle was introduced into the center of the tumor; then, 60 W of the radiofrequency energy was delivered by the generator with an 8-minute duration for every single energy application.
  Arms: RFA group
Procedure: hepatic resection — SR was carried out under general anesthesia using a right subcostal incision with a midline extension.Intra-operative ultrasonography was performed routinely to evaluate the tumor burden, liver remnant, and the possibility of a negative resection margin. Anatomic resection, in the form of segmentectomy and/or subsegmentectomy as described by Makuuchi et al. (16) was the preferred surgical method of liver resection. Pringle's maneuver was routinely used with a clamp and unclamp time of 10 min and 5 min, respectively; this technique was used repeatedly throughout the entire procedure. Hemostasis of the raw liver surface was done with suturing and application of fibrin glue.
  Arms: HR group

SUMMARY:
Recently, a clinical trial has shown that PRFA is as effective as HR for small HCC in terms of overall survival and disease-free survival. This has prompted some authors to suggest that PRFA could be more suitable than HR for early stage HCC. Some authors also have suggested that PRFA can be considered the treatment of choice for patients with single HCC ≤ 2.0 cm, even when HR is possible. On the other hand, some tumors (subcapsular location, adjacent to intestinal loops or main bile ducts) may be unsuitable for PRFA because of the risk of bleeding, tumor seeding, bile leakage, perforation, and so on. Furthermore, in our previous experience, some tumors (with deep locations, which were included as "central HCC") may be also unsuitable for HR because of risks of more injury of normal liver tissue, blood loss after resection, and so on. Therefore, the appropriate therapeutic option for these HCC tumors ≤ 2 cm, especially for central HCC, is still under debate. To clarify this issue, the investigators conducted a study that included a consecutive series of patients with single resectable HCC < 2.0 cm in diameter, who underwent PRFA or HR.

DETAILED DESCRIPTION:
With the development of medical science, more and more patients are being diagnosed with hepatocellular carcinoma (HCC) at an early stage (single ≤ 5 cm in diameter or ≤ 3 nodules, ≤ 3 cm in diameter) allowing for radical treatment by hepatic resection (HR), liver transplantation, or percutaneous ablation . Liver transplantation can eliminate the tumor and cirrhosis at the same time, and is considered to be the most appropriate treatment for these patients. However, the lack of liver donors is a major limitation. Until now, HR has still been considered as the first-choice treatment for these patients, which may offer a 5-year survival rate above 50%. Percutaneous ablation, including percutaneous ethanol injection (PEI) and percutaneous radiofrequency ablation (PRFA), is usually considered to be a second-choice treatment for small HCC which is unresectable due to impaired liver function, and liver transplantation is not indicated.

Recently, a clinical trial has shown that PRFA is as effective as HR for small HCC in terms of overall survival and disease-free survival. This has prompted some authors to suggest that PRFA could be more suitable than HR for early stage HCC. Some authors also have suggested that PRFA can be considered the treatment of choice for patients with single HCC ≤ 2.0 cm, even when HR is possible. On the other hand, some tumors (subcapsular location, adjacent to intestinal loops or main bile ducts) may be unsuitable for PRFA because of the risk of bleeding, tumor seeding, bile leakage, perforation, and so on. Furthermore, in our previous experience, some tumors (with deep locations, which were included as "central HCC") may be also unsuitable for HR because of risks of more injury of normal liver tissue, blood loss after resection, and so on. Therefore, the appropriate therapeutic option for these HCC tumors ≤ 2 cm, especially for central HCC, is still under debate. To clarify this issue, the investigators conducted a study that included a consecutive series of patients with single resectable HCC < 2.0 cm in diameter, who underwent PRFA or HR.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 - 75 years, who refused liver transplantation;
2. presence of solitary HCC measuring ≤ 2.0 cm in diameter;
3. resectable disease, which is defined as the possibility of completely removing all tumors and retaining a sufficient liver remnant to maintain liver function, as assessed by our surgery team;
4. Eastern Co-operative Oncology Group performance (ECOG) status 0 (15);

Exclusion Criteria:

1. severe coagulation disorders (prothrombin activity < 40% or a platelet count of < 40,000 / mm3;
2. the presence of vascular invasion or extrahepatic spread on imaging;
3. Child-Pugh class C liver cirrhosis or evidence of hepatic decompensation including ascites, esophageal or gastric variceal bleeding, or hepatic encephalopathy;
4. previous treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 year

SECONDARY OUTCOMES:
disease-free survival | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: min-shan chen, Ph.D.,M.D., Principal Investigator — Cancer Center, Sun Yat-set University
Locations (1):
- Cancer Center, Sun Yat-set University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chen MS, Li JQ, Zheng Y, Guo RP, Liang HH, Zhang YQ, Lin XJ, Lau WY. A prospective randomized trial comparing percutaneous local ablative therapy and partial hepatectomy for small hepatocellular carcinoma. Ann Surg. 2006 Mar;243(3):321-8. doi: 10.1097/01.sla.0000201480.65519.b8. PMID 16495695